CLINICAL TRIAL: NCT06378788
Title: Ultrasound-imaged Muscle Architecture and Muscle Strength in Fibromyalgia and it's Correlation With Pain, Disease Activity, and Functionality
Brief Title: Muscle Architecture and Muscle Strength in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/211
Record Dates: First submitted 2024-04-04; First posted 2024-04-22 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia; Sarcopenia; Muscle Weakness
Keywords: muscle strength; musculoskeletal ultrasound
MeSH Terms: conditions — Fibromyalgia; Sarcopenia; Muscle Weakness | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: Patients meeting the diagnostic criteria of 2016 American College of Rheumatology (ACR) guide for fibromyalgia
  Interventions: Other: Demographic information form; Diagnostic Test: widespread pain index (WPI); Diagnostic Test: symptom severity scale (SSS); Diagnostic Test: Fibromyalgia Impact Questionnaire (FIQ); Diagnostic Test: Tender Point examination; Other: Muscle Architecture visualized with ultrasound; Other: Sarcopenia assessed by measuring isometric strengths of different parts of the body; Other: Timed Up & Go (TUG)
- Control: healthy participants
  Interventions: Other: Demographic information form; Other: Muscle Architecture visualized with ultrasound; Other: Sarcopenia assessed by measuring isometric strengths of different parts of the body

INTERVENTIONS:
Other: Demographic information form — aims to collect basic demographic data( Age reported by years , weight and height will be combined to report Body Mass index (BMİ) in kg/m2, Smoking habit reported as smoker or non-smoker , Level of Education reported as illiterate, literate, Primary school, Middle school, High school, University or Post-graduate, Profession type, Significant medical records and Medications.
Diagnostic Test: widespread pain index (WPI) — The Widespread Pain Index is a 19-point checklist that assesses the presence of pain or tenderness (within the prior seven days) in 19 specific areas of the body; each affected area receives one point. The 19 regions on the WPI include the following:
  Right and left jaw, Right and left shoulder girdle, Right and left upper arm, Right and left lower arm, Right and left hip/buttock Right and left upper leg Right and left lower leg Upper and lower back Neck Chest Abdomen A fibromyalgia diagnosis is confirmed if a WPI is ≥7 with an SS scale ≥5 OR a WPI range between 4-6 with an SS scale ≥ 9.
  Groups: Fibromyalgia
Diagnostic Test: symptom severity scale (SSS) — SS scale score: Fatigue, waking unrefreshed, and cognitive symptoms. For each of the three symptoms above, indicate the severity level over the past week utilizing the following scale: 0 no problem; 1 slight or mild problems, generally mild or intermittent; 2 moderate, considerable problems, often present and/or at a moderate level; 3 severe: pervasive, continuous, life-disturbing problems. Considering somatic symptoms in general, indicate whether the patient has: 0 for no symptoms, 1 for a few symptoms, 2 for a moderate number of symptoms, and 3 for many symptoms. The SS scale score sums the severity of the 3 symptoms (fatigue, waking unrefreshed, cognitive symptoms) plus the severity) of general somatic symptoms. The final score is between 0 and 12.
  Groups: Fibromyalgia
Diagnostic Test: Fibromyalgia Impact Questionnaire (FIQ) — The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. The FIQ is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression.
  Groups: Fibromyalgia
Diagnostic Test: Tender Point examination — Tender points are specific sites on the body that cause pain when pressed.. There are 9 pairs of tender points. Each pair has one point on each side of the body, for a total of 18 points.Prior to 2010, the diagnosis of fibromyalgia required at least 11 painful point of 18 but now tender points are no longer used as a diagnostic tool. The score will be reported as the number of tender points found with palpation.
  Groups: Fibromyalgia
Other: Muscle Architecture visualized with ultrasound — The three head of Quadratus femoris ( Vastus lateralis, Vastus Medialis and Rectus Femoris), Tibialis Anterior, the two heads of Gastrocnemius ( vastus Lateralis and vastus Medialis) ultrasonography will be performed to evaluate muscle thickness, pennation angle and fascicle length.
Other: Sarcopenia assessed by measuring isometric strengths of different parts of the body — Cervical Flexion (CF), Cervical Extension (CE), Right and Left Cervical Lateral Flexion (CLF R/L), Truncal flexion (TF), Truncal extension (TE), Shoulder flexion (SF), Shoulder extension (SE), Shoulder abduction (SAB), Shoulder internal rotation (SIR) and Shoulder external rotation (SER), Hip flexion (HF), Hip extension (HE), hip abduction (HAB), hip internal rotation (HIR), hip external rotation (HER), knee extension (KE), Knee Flexion (KF), Ankle Dorsiflexion (ADF) and Ankle Plantar flexion (APF) muscle strengths will be evaluated with hand held dynamometer
Other: Timed Up & Go (TUG) — The test will be used by investigators as a simple evaluative test used to measure participants functional mobility.
  Groups: Fibromyalgia

SUMMARY:
The goal of this observational study is to determine whether there is decrease in muscle mass and muscle strength in Fibromyalgia Syndrome (FMS) patients in comparison to controls. And to determine whether these parameters are correlated with clinical ones. Briefly the main questions investigators aims to answer are:

* Is there a significant difference in muscle morphology between FMS and controls?
* Is there a significant difference in muscle strength between FMS and controls?
* Is there a relationship between muscle thickness and pennation angle of the Quadriceps, gastrocnemius medialis, gastrocnemius lateralis and Tibialis anterior muscles and disease activity, pain and functionality?
* Is there a correlation between muscle strength in FMS and disease activity, pain and functionality?

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) was named by Smythe and Moldofsky when they defined tender points in 1970s. It is defined as chronic, generalized musculoskeletal pain accompanying with fatigue, sleep disturbance , cognitive and somatic disturbance. FMS has variable prevalence as %0,7-11 and usually affects middle aged women. It is second most common rheumatologic disease after osteoarthritis and thought to be the most common reason for musculoskeletal pain in middle aged women.

Recent studies have reported that both sarcopenia and decreased muscle strength occur in patients with chronic inflammatory diseases such as rheumatoid arthritis. There are concerns that sarcopenia may affect exercise tolerance, activities of daily living, and ultimately have a negative impact on cardiovascular fitness and physical and emotional well-being. On the other hand there is researches that support inflammation-driven pathways in the pathogenesis of fibromyalgia. Given the risk of pain related reduction in physical activity, patients are expected to have accelerated muscle wasting , decreased muscle strength and endurance and functionality.

However, there is no study that focused on muscle architecture and strength in FMS. This led us to design our study which will evaluate patients lower extremity muscles' thickness and pennation angles by ultrasound , most daily used muscles' strength by dynamometer, functionality by timed-up test and try to find whether there is a correlation between these parameters and patients' disease activity which will be determined with FMS specific scales.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the 2016 ACR (American College of Rheumatology) diagnostic criteria.
* Diagnosed at least 1 year ago.

Exclusion Criteria:

* Patients diagnosed with other rheumatological diseases, muscle diseases, or neuropathies.
* Patients with a history of trauma affecting muscle morphology.
* Patients engaging in regular exercise (at least 3-4 times a week for a minimum of 40 minutes).
* Patients with uncontrolled comorbid diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fisrt group: Fibromyalgia diagnosed patient group Second group: Healthy control group
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Quadriceps Femoris Vastus Lateralis Muscle Thickness | through study completion, an average of 16 weeks
  Vastus lateralis ultrasonography will be performed to evaluate muscle thickness.
Quadriceps Femoris Vastus Lateralis Fascicle Length | through study completion, an average of 16 weeks
  Vastus lateralis ultrasonography will be performed to evaluate fascicle length through measuring pennation angle (PA).
Quadriceps Femoris Vastus Medialis Muscle Thickness | through study completion, an average of 16 weeks
  Vastus Medialis ultrasonography will be performed to evaluate muscle thickness.
Quadriceps Femoris Vastus Medialis Fascicle Length | through study completion, an average of 16 weeks
  Vastus Medialis ultrasonography will be performed to evaluate fascicle length through measuring pennation angle (PA).
Quadriceps Femoris Rectus Femoris Muscle Thickness | through study completion, an average of 16 weeks
  Rectus Femoris ultrasonography will be performed to evaluate muscle thickness.
Quadriceps Femoris Rectus Femoris Fascicle Length | through study completion, an average of 16 weeks
  Rectus Femoris ultrasonography will be performed to evaluate fascicle length through measuring pennation angle (PA).
Tibialis Anterior Muscle Thickness | through study completion, an average of 16 weeks
  Tibialis Anterior ultrasonography will be performed to evaluate muscle thickness.
Tibialis Anterior Muscle Fascicle Length | through study completion, an average of 16 weeks
  Tibialis Anterior ultrasonography will be performed to evaluate fascicle length through measuring pennation angle (PA).
Gastrocnemius Muscle Vastus Medialis Muscle Thickness | through study completion, an average of 16 weeks
  Gastrocnemius muscle vastus medialis ultrasonography will be performed to evaluate muscle thickness.
Gastrocnemius Muscle Vastus Medialis Fascicle Length | through study completion, an average of 16 weeks
  Gastrocnemius muscle vastus medialis ultrasonography will be performed to evaluate fascicle length through measuring pennation angle (PA).
Gastrocnemius Muscle Vastus Lateralis Muscle Thickness | through study completion, an average of 16 weeks
  Gastrocnemius muscle vastus lateralis ultrasonography will be performed to evaluate muscle thickness.
Gastrocnemius Muscle Vastus Lateralis Fascicle Length | through study completion, an average of 16 weeks
  Gastrocnemius muscle vastus lateralis ultrasonography will be performed to evaluate fascicle length through measuring pennation angle (PA).
Cervical Muscle strength | through study completion, an average of 16 weeks
  Isometric Cervical Flexion (CF), Isometric Cervical Extension (CE) and Right and Left Isometric Cervical Lateral Flexion (CLF R/L) strengths will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Truncal Muscle strength | through study completion, an average of 16 weeks
  Isometric Truncal flexion (TF)and Isometric Truncal extension (TE) strengths will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Shoulder Muscle strength | through study completion, an average of 16 weeks
  Isometric Shoulder flexion (SF), Isometric Shoulder extension (SE), Isometric Shoulder abduction (SAB), Isometric Shoulder internal rotation (SIR) and Isometric Shoulder external rotation (SER) strengths will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Hip Muscle strength | through study completion, an average of 16 weeks
  Isometric Hip flexion (HF), Isometric Hip extension (HE), Isometric Hip abduction (HAB), Isometric Hip internal rotation (HIR) and Isometric Hip external rotation (HER), strengths will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Knee Muscle strength | through study completion, an average of 16 weeks
  Isometric Knee extension (KE) and Isometric Knee Flexion (KF) strengths will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Ankle Muscle strength | through study completion, an average of 16 weeks
  Isometric Ankle Dorsiflexion (ADF) and Isometric Ankle Plantar flexion (APF) strengths will be calculated with hand-held dynamometer(Lafayette Manual Muscle Tester ) and reported as kilograms.
Timed Up & Go (TUG) | through study completion, an average of 16 weeks
  The patient sits in the chair with his/her back against the chair back. On the command "go," the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down.
  Timing begins at the instruction "go" and stops when the patient is seated and will be reported by seconds.
  This test aim to determine patients functional state and mobility .

CONTACTS AND LOCATIONS:
Overall Officials: Delal Ozturk, Res.Ass, Principal Investigator — Bezmialem VU
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Privacy reasons

REFERENCES:
- [Background] Gyorfi M, Rupp A, Abd-Elsayed A. Fibromyalgia Pathophysiology. Biomedicines. 2022 Nov 29;10(12):3070. doi: 10.3390/biomedicines10123070. PMID 36551826
- [Background] Blanco I, Beritze N, Arguelles M, Carcaba V, Fernandez F, Janciauskiene S, Oikonomopoulou K, de Serres FJ, Fernandez-Bustillo E, Hollenberg MD. Abnormal overexpression of mastocytes in skin biopsies of fibromyalgia patients. Clin Rheumatol. 2010 Dec;29(12):1403-12. doi: 10.1007/s10067-010-1474-7. Epub 2010 Apr 30. PMID 20428906
- [Background] Ruggiero L, Manganelli F, Santoro L. Muscle pain syndromes and fibromyalgia: the role of muscle biopsy. Curr Opin Support Palliat Care. 2018 Sep;12(3):382-387. doi: 10.1097/SPC.0000000000000355. PMID 29912728
- [Background] Chinn S, Caldwell W, Gritsenko K. Fibromyalgia Pathogenesis and Treatment Options Update. Curr Pain Headache Rep. 2016 Apr;20(4):25. doi: 10.1007/s11916-016-0556-x. PMID 26922414
- [Background] Lund N, Bengtsson A, Thorborg P. Muscle tissue oxygen pressure in primary fibromyalgia. Scand J Rheumatol. 1986;15(2):165-73. doi: 10.3109/03009748609102084. PMID 3462905
- [Background] Thieme K, Rose U, Pinkpank T, Spies C, Turk DC, Flor H. Psychophysiological responses in patients with fibromyalgia syndrome. J Psychosom Res. 2006 Nov;61(5):671-9. doi: 10.1016/j.jpsychores.2006.07.004. PMID 17084146
- [Background] Zetterman T, Markkula R, Partanen JV, Miettinen T, Estlander AM, Kalso E. Muscle activity and acute stress in fibromyalgia. BMC Musculoskelet Disord. 2021 Feb 14;22(1):183. doi: 10.1186/s12891-021-04013-1. PMID 33583408
- [Background] Larsson A, Palstam A, Bjersing J, Lofgren M, Ernberg M, Kosek E, Gerdle B, Mannerkorpi K. Controlled, cross-sectional, multi-center study of physical capacity and associated factors in women with fibromyalgia. BMC Musculoskelet Disord. 2018 Apr 19;19(1):121. doi: 10.1186/s12891-018-2047-1. PMID 29673356
- [Background] Cigaran-Mendez M, Ubeda-D'Ocasar E, Arias-Buria JL, Fernandez-de-Las-Penas C, Gallego-Sendarrubias GM, Valera-Calero JA. The hand grip force test as a measure of physical function in women with fibromyalgia. Sci Rep. 2022 Mar 1;12(1):3414. doi: 10.1038/s41598-022-07480-1. PMID 35233066
- [Background] Kuzu O, Aras B. Sonographic measurement of the neck extensor muscle thickness in patients with fibromyalgia. Musculoskelet Sci Pract. 2022 Jun;59:102541. doi: 10.1016/j.msksp.2022.102541. Epub 2022 Feb 26. PMID 35240562
- [Background] Blazevich AJ, Gill ND, Zhou S. Intra- and intermuscular variation in human quadriceps femoris architecture assessed in vivo. J Anat. 2006 Sep;209(3):289-310. doi: 10.1111/j.1469-7580.2006.00619.x. PMID 16928199
- [Background] Yurdakul OV, Ince OE, Bagcier F, Kara M, Kultur E, Aydin T. Evaluating the strength of spinal and proximal girdle muscles in patients with axial spondyloarthritis: Correlation with activity, disability, and functionality. Int J Rheum Dis. 2021 May;24(5):701-710. doi: 10.1111/1756-185X.14102. Epub 2021 Mar 22. PMID 33750032